CLINICAL TRIAL: NCT06135506
Title: Artificial Intelligence-Assisted/Computer Guided Ridge Splitting for the Treatment of Horizontal Ridge Defects With Simultaneous Guided Implant Placement: Randomized Controlled Clinical Study
Brief Title: Artificial Intelligence/Computer Guided Ridge Splitting for Treating Horizontal Ridge Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Walid Elamrousy, Assistant Professor of periodontology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-74
Record Dates: First submitted 2023-11-11; First posted 2023-11-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Alveolar Bone Resorption; Dental Implant Failure Nos
Keywords: Artificial intelligence; ridge splitting; computer-guided surgery

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): conventional ridge splitting with conventional simultaneous implant placement.
  Interventions: Procedure: free-hand ridge splitting
- study group (Experimental): computer guided ridge splitting assisted by artificial intelligence with simultaneous computer guided implant placement.
  Interventions: Procedure: AI/guided ridge splitting

INTERVENTIONS:
Procedure: free-hand ridge splitting — Midcrestal incision will be followed by reflection of full thickness flap. Midcrestal cut without vertical osteotomy will be done using piezosurgery unit, and then the cut will be extended deep to the implant length. The ridge will be expanded progressively using bone wedges. Dental implant fixtures will be placed stably with 1 mm minimal thickness of buccal bone plate. Surgical site will be completely closed, and wound edges will be sutured in a tension-free way.
  Arms: control group
Procedure: AI/guided ridge splitting — The patient specific guides will be placed and fixed by monocortical osteosynthesis screws at the pre-planned positions at the labial buccal mucosa.
  A midcrestal cut will be performed on the crest of alveolar ridge guided by the guide slits. The cuts will be expanded progressively using bone wedges through the guide slits gradually lateralize and expand the labial alveolar plate of bone, so the labial cortex will move through the intentionally created micro gap till it touches the fitting aspect of the patient specific guide. Implant drills will be inserted through the guiding holes in the surgical guide and the implant osteotomy sites will be prepared. Finally, implants will be inserted in the osteotomy sites using torque-wrench in a self-tapping fashion engaging palatal and basal bone for primary stability.
  Arms: study group

SUMMARY:
Aim of the current randomized clinical trial is to evaluate and compare the effectiveness of computer-guided ridge splitting approach assisted by artificial intelligence versus conventional approach combined with simultaneous implant Placement.

DETAILED DESCRIPTION:
Ridge split technique is considered one of the successful horizontal bone augmentation procedures especially in maxilla for the management of horizontal ridge defects. This was adapted by Summers in 1994.

Guided implant surgery was used in dental implant surgery to achieve accuracy and an overall predictability. Successful guided implant workflow depends on 3-dimensional image acquisition and precise model fabrication.

Artificial intelligence application in implant dentistry has ushered in a new era of precision and efficiency demonstrating improved implant survival rates and patient satisfaction and enhance the integration of technologies with digital workflows.

ELIGIBILITY:
Inclusion Criteria:

* The target population with inadequate bone volume for implant placement due to width insufficiency of maxillary anterior alveolar ridges.
* Age ranges from 25-40 years of both sexes.
* No gender restrictions were considered for initial screening.
* Absence of any complicating systemic condition that may contraindicate surgical procedures and implant placement.
* Adequate oral hygiene.
* Eligible participants should present good general health and agree to random assignment to any of the two parallel study groups.
* Participants had minimum 3 months as post extraction healing period and horizontal maxillary anterior ridge defects with at least bone width of 3 mm and bone height of 13 mm.

Exclusion Criteria:

* Vertical ridge defect.
* Undercut on the labial/buccal side.
* Thick cortical bone without cancellous bone inside.
* Uncontrolled systematic disorders as, diabetes mellitus, uncontrolled periodontal disease, history of head and neck radiotherapy, smokers, pregnancy, noncompliant patients, allergy to the used medications, uncooperative individuals or those unable to attend the study follow-up appointments.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-19 (Actual)

PRIMARY OUTCOMES:
alveolar ridge width | 9-month.
  CBCT will have taken immediately after surgery, at 6 and 9 months postoperatively to evaluate ridge width using OnDemand3D™ App-3D CBCT software.
  The alveolar ridge width will be measured buccolingually in axial view 2 mm apical to the implant collar margin.

SECONDARY OUTCOMES:
vertical bone height | 9-months
  CBCT will have taken immediately after surgery, at 6 and 9 months postoperatively to evaluate vertical bone height.
  Mesiodistal vertical bone height will be measured using coronal view from a fixed anatomical landmark point to the mesial and distal marginal bone level. Moreover, sagittal view will be used to measure buccolingual vertical bone height extending from fixed anatomical reference point to the buccal and lingual alveolar crest. usinng CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Walid Elamrousy, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided